CLINICAL TRIAL: NCT02784639
Title: Comparison of KRAS/BRAF Mutational Status Between Tumor Tissue Section Analysis With Conventional Techniques and Plasma Samples Analysis (KPLEX2)
Brief Title: Comparison of KRAS/BRAF Mutational Status With Conventional Techniques and Plasma Samples Analysis
Acronym: KPLEX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICM2013/08
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
Keywords: KRAS/BRAF mutational status
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- determination of KRAS mutation (Other): circulating cell free DNA (ccfDNA) plasma analysis
  Interventions: Other: Plasma Analysis of circulating cell free DNA; Other: Tumor tissue analysis of circulating cell free DNA

INTERVENTIONS:
Other: Plasma Analysis of circulating cell free DNA
Other: Tumor tissue analysis of circulating cell free DNA

SUMMARY:
The goal of this multicenter prospective study is to validate, and ultimately translate in routine clinical practice, the use of plasma analysis of ccfDNA for the determination of KRAS mutation status in mCRC patients.

DETAILED DESCRIPTION:
Analyzing qualitatively and quantitatively genetic alterations with an efficient, simple and cost-effective test from blood samples could optimize therapeutic decision-making and personalized cancer care. Cell-free DNA (ccfDNA) levels in the plasma of CRC patients are significantly higher than in healthy patients. These levels decrease progressively in tumor-free patients during the follow-up period and increase in patients with recurrence or metastasis. In the near future, the detection of circulating DNA (ccfDNA) could therefore represent a technology breakthrough for diagnosis, prognosis, detection of tumor growth and cancer patient follow up.

We designed a refined and innovative method which simultaneously allows the determination of three parameters: the specific quantification of tumor-derived ccfDNA, the ccfDNA fragmentation index, and SNP (Single Nucleotide Polymorphism) or point mutation detection. In addition to its unprecedented sensitivity and specificity, this qPCR based-method (termed IntPlex®), recently patented by the CNRS, is easy and rapid, and the first multiplexed test for ccfDNA.

Evaluation and validation of the IntPlex® test was examined in response to the pressing need to determine the KRAS/BRAF mutational status before anti-EGFR therapy in CRC patients. As a consequence, the method was adapted to detect the six more frequent KRAS mutations in CRC (G12D, G12V, G13D, G12S, G12C, G12A) and the BRAF V600E. We then carried out the first blinded prospective study to compare KRAS and BRAF mutational status data obtained from the analysis of tumor tissue by routine gold standard methods and of plasma DNA using our original method (ASCO oral communication). The mutational status was determined by both methods in 70 patient samples. Our results clearly showed for the first time that ccfDNA analysis for KRAS mutation could replace advantageously tumor-section analysis. CcfDNA analysis showed 100% specificity and sensitivity for the BRAF V600E mutation. For the six tested KRAS point mutations, the method exhibited 100% specificity and 87% sensitivity with a concordance value of 96%.

The goal of this multicenter prospective study is to validate, and ultimately translate in routine clinical practice, the use of plasma analysis of ccfDNA for the determination of KRAS mutation status in mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of colorectal cancer

* Synchronous or metachronous metastatic colorectal cancer
* Patient for whom the KRAS status is requested for therapeutic decision-making
* Male or female ≥ 18 years old
* Patients must be affiliated to a Social Security System
* Patient information and written informed consent form signed prior to any study specific procedures

Exclusion Criteria:

* History of other malignancy within the previous 5 years (except for appropriately treated carcinoma in situ of the cervix and non-melanoma skin carcinoma)
* Blood transfusion within 1 week prior to blood collection
* Patients having received any chemotherapy or/and radiotherapy within 15 days prior to blood collection
* Patients with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Area under ROC curve | 12 month
  Area under the ROC curve of the mutation percentage obtained from plasma ccfDNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: MARC YCHOU, Principal Investigator — Institut régional du Cancer de Montpellier

IPD SHARING:
Plan to Share IPD: No